CLINICAL TRIAL: NCT00918827
Title: Study of Biomarkers in Tissue Samples of Patients With Stage III Colon Cancer Treated With Adjuvant Chemotherapy Comprising Fluorouracil-Based Regimens(B-CAST)
Brief Title: Study of Tumor Samples From Patients With Stage III Colon Cancer Who Have Undergone Surgery and Chemotherapy
Status: Completed | Type: Observational
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Tokyo Medical and Dental University (Other)
Responsible Party: Sponsor
Other Study IDs: CDR0000642386; TMDU-TRICC0807 (Other: National Cancer Institute); UMIN000002013 (Registry Identifier: UMIN-CTR)
Record Dates: First submitted 2009-06-09; First posted 2009-06-11 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-06

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the colon; stage III colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
RATIONALE: Studying samples of tumor tissue in the laboratory from patients with cancer who have undergone surgery and chemotherapy may help doctors predict how well patients will respond to treatment.

PURPOSE: This research study is looking at tumor samples from patients with stage III colon cancer who have undergone surgery and chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Identify predictive factors of efficacy and safety of adjuvant chemotherapy comprising fluorouracil-based regimens in patients with stage III colon cancer.
* Investigate possibility of "personalized treatment" with adjuvant chemotherapy based on the predictive factors identified.

OUTLINE: Patients' tumor tissue samples are collected for protein expression levels of thymidine phosphorylase (TP), dihydropyrimidine dehydrogenase (DPD), VEGF, EGFR, mRNA-expression levels of TP, DPD, thymidylate synthase (TS), and orotate phosphoribosyl transferase (OPRT) by ELISA, Human Duo Set, and RT-PCR assays.

Patients' enzyme expression levels are compared with their clinical data.

ELIGIBILITY:
<Inclusion criteria>

* Pathologically confirmed stage III colon adenocarcinoma
* Curatively resected (R0)
* Patients scheduled for treatment with fluorouracil-based post-operative adjuvant chemotherapy
* Provided written informed consent

<Exclusion criteria>

* Synchronous or metachronous multiple cancers
* Contraindications for fluorouracil-based chemotherapy
* Patients who have initiated neo-adjuvant chemotherapy or radiotherapy prior to participating in this study
* Ineligible patients according to the investigator's judgement

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pathologically confirmed stage III colon adenocarcinoma patients who are given treatment with fluorouracil-based post-opeartive adjuvant chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 2128 (Actual)
Dates: Start 2009-04-01; Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Relationship between expression levels of enzymes and disease-free survival, relapse-free survival, and overall survival | 5 years after the end of registration
Relationship between expression levels of enzymes and adverse effects | 5 years after the end of registration
Disease-free survival | Until the day on which an event reveals during the 5 year observational period
Relapse-free survival | Until the day on which an event reveals during the 5 year observational period

CONTACTS AND LOCATIONS:
Overall Officials: Kenichi Sugihara, MD, PhD, Principal Investigator — Tokyo Medical and Dental University
Locations (1):
- Tokyo Medical and Dental University, Tokyo, Japan

REFERENCES:
- [Derived] Ishiguro M, Kotake K, Nishimura G, Tomita N, Ichikawa W, Takahashi K, Watanabe T, Furuhata T, Kondo K, Mori M, Kakeji Y, Kanazawa A, Kobayashi M, Okajima M, Hyodo I, Miyakoda K, Sugihara K. Study protocol of the B-CAST study: a multicenter, prospective cohort study investigating the tumor biomarkers in adjuvant chemotherapy for stage III colon cancer. BMC Cancer. 2013 Mar 25;13:149. doi: 10.1186/1471-2407-13-149. PMID 23530572